CLINICAL TRIAL: NCT05695456
Title: Targeted Elimination Diet in EoE Patients Following Identification of Trigger Nutrients Using Confocal Laser Endomicroscopy
Acronym: CLE-EoE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: S66223
Record Dates: First submitted 2022-03-15; First posted 2023-01-25 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-03

CONDITIONS: Eosinophilic Esophagitis
Keywords: confocal laser endomicroscopy; 6-food elimination diet; personalized exclusion diet
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Intervention Model Description: A double-blind cross-over dietary elimination study: Patients with a positive CLE reaction to one or two specific nutrients will then be randomized to a blinded exclusion diet for 6 weeks of those nutrients or to exclusion of another tested nutrient that yielded no change in CLE (=sham diet), in a cross-over fashion. Patients with no CLE reaction will undergo an empirical exclusion diet of gluten-containing grains for 6 weeks. To mirror the crossover character of the intervention, CLE negative patients will then undergo a milk exclusion diet for 6 weeks (order is interchangeable).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Nor the participant, nor the primary or secondary investigators involved in the study will know to which nutrients the patient reacted as assessed by CLE, nor will they know what the order of the diet is (sham or real). An investigator who did not participate in the CLE will give dietary instructions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CLE positive patients real/sham (Active Comparator): In this arm, participants who reacted to one or two nutrients during CLE will follow a personalized exclusion diet consistent of the nutrient to which they reacted, after which they will follow a sham diet in a blinded cross-over fashion.
  Interventions: Other: personalized exclusion diet based on CLE
- CLE positive patients sham/real (Sham Comparator): In this arm, participants who reacted to one or two nutrients during CLE will follow a sham diet for 6 weeks, and than a personalized exclusion diet consistent of the nutrient to which they reacted, in a blinded cross-over fashion.
  Interventions: Other: personalized exclusion diet based on CLE
- CLE negative patients (Sham Comparator): In this arm, participants who did not react to one of the nutrients during CLE will follow a control diet consistent of milk exclusion for 6 weeks, after which they will follow a gluten exclusion diet for 6 weeks, or the other way around.
  Interventions: Other: empiric exclusion diet

INTERVENTIONS:
Other: personalized exclusion diet based on CLE — personalized exclusion diet based on CLE
  Arms: CLE positive patients real/sham; CLE positive patients sham/real
Other: empiric exclusion diet — exclusion diet with milk or gluten-containing grains
  Arms: CLE negative patients

SUMMARY:
Using confocal laser endomicroscopy (CLE), gastrointestinal allergic reactions to certain foods in the duodenum will be evaluated on a cellular level. After that, a personalized exclusion diet will be followed based on the CLE results for 6 weeks, sham-controlled, in a cross-over fashion. Gastroscopy with esophageal biopsies will be repeated after each diet.

DETAILED DESCRIPTION:
Eosinophilic esophagitis is an antigen driven esophagitis, that is characterized by symptoms of dysphagia often leading to food impaction, and that leads to strictures and esophageal motility disorders, with a significant impact on quality of life. Current treatment options include proton pump inhibitors (PPI's) and topical steroids, and also the empiric 6-food elimination diet (6FED). In this diet, the 6 most frequently implicated foods are excluded and reintroduced one by one (milk, gluten containing grains, egg, soy, nuts, fish & shellfish). However, this is a complicated and long process, including several endoscopies with esophageal biopsies.

Confocal laser endomicroscopy (CLE) is a technique that allows to detect gastrointestinal allergic reactions in the duodenum, and to visualize them on a molecular level in real-time. The CLE probe is passed through the working channel of a standard gastroscope, up against the duodenal mucosa. After intravenous injection of fluorescein as contrast medium, the duodenal epithelium is visualized on a cellular level, including food protein mediated extravasation of fluorescein into the lumen. The 6 foods of the 6FED are sprayed on the epithelium one by one, after which a reaction is awaited. Previous use of CLE has shown that more than half of Eosinophilic esophagitis (EoE) patients reacts to one or more foods during CLE.

In this double blind randomized cross-over study the effect a personalized elimination diet, based on the reaction during CLE, is compared to a sham diet, in patients with eosinophilic esophagitis, and insufficient response or intolerance to PPI's. Both diets will be followed for 6 weeks, after which gastroscopy with esophageal biopsies will be repeated. Patients that do not have a reaction to the 6 foods will act as controls, following a control diet with milk and gluten in a cross-over fashion.

ELIGIBILITY:
Inclusion Criteria:

* Eosinophilic Esophagitis, with peak eosinophil count of >15 eos/HPF and symptoms of dysphagia at least 2 days per week
* Patients have had a trial of high-dose PPI for at least 8 weeks, with either documented non-response or intolerance to the medication
* Patients aged between 18 and 70 years old
* Signed written informed consent
* Eosinophilic Esophagitis, with peak eosinophil count of >15 eos/HPF and symptoms of dysphagia at least 2 days per week
* Patients have had a trial of high-dose PPI for at least 8 weeks, with either documented non-response or intolerance to the medication
* Patients aged between 18 and 70 years old
* Signed written informed consent

Exclusion criteria:

* IgE-mediated food anaphylaxis for 1 of the trigger nutrients
* History of major gastrointestinal surgery complicating esophago-gastro-duodenoscopy
* Gastro-esophageal reflux disease (GERD) Los Angeles grade C or D
* Esophageal strictures, too narrow to pass with a normal gastroscope
* Endoscopic dilation in the esophagus in the 4 weeks prior to inclusion
* Celiac disease
* Recent use (within two weeks) of non-steroidal anti-inflammatory drugs (NSAIDs), systemic histamine-receptor antagonists, mast cell stabilizers, opioids.
* Proton pump inhibitors must be either stopped for at least 4 weeks, or continued on a stable dosage throughout the study period.
* Corticosteroids should be stopped for at least 4 weeks.
* Allergy to fluorescein, Xylocain or Propofol
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difference in response | 2 years
  Difference in response (defined as normalization of peak eosinophil count in esophageal mucosal biopsies <15 eosinophils/HPF) in patients undergoing duodenal CLE-targeted elimination diet compared to the sham diet

SECONDARY OUTCOMES:
Further histological outcomes | 2 years
  Difference in deep remission (defined as reduction of peak eosinophil count <6 eosinophils/HPF) before and after the targeted elimination diet respectively, compared with the sham diet
Further histological outcomes | 2 years
  Difference in peak eosinophil count (eosinophils/HPF) before and after the targeted elimination diet, compared with the sham diet
Symptomatic changes in patients undergoing duodenal CLE-targeted elimination diet compared to the sham diet | 2 years
  difference in symptoms using the DSQ (dysphagia symptom questionnaire), with a score from 0 (meaning no symptoms) to 10 (worse outcome).
endoscopic changes in patients undergoing duodenal CLE-targeted elimination diet compared to the sham diet | 2 years
  Difference in endoscopic reference score (EREFS) ranging from E0R0E0F0S0 (no endoscopic abnormalities) to E2R2E2F2S2 (worse endoscopic features)
change in esophageal and duodenal permeability parameters 1 | 2 years
  using ussing chamber experiments, where human biopsies our mounted in between two chambers, and the transepithelial electrical resistance (TEER) is measured across the chambers
change in esophageal and duodenal permeability parameters 2 | 2 years
  using ussing chamber experiments, where human biopsies our mounted in between two chambers, and the transepithelial flux of a high molecular weight protein is measured by labeling the molecule with a fluorescent dye.
Baseline and post-exposure duodenal mast cell and eosinophil counts on histology | 2 years
  Baseline and post-exposure duodenal mast cell and eosinophil counts on histology
Differences in duodenal permeability measures in CLE positive, CLE negative EoE patients and healthy controls before and after nutrient application 1 | 2 years
  using ussing chamber experiments, where human biopsies our mounted in between two chambers, and the transepithelial electrical resistance (TEER) is measured across the chambers
Differences in duodenal permeability measures in CLE positive, CLE negative EoE patients and healthy controls before and after nutrient application 2 | 2 years
  using ussing chamber experiments, where human biopsies our mounted in between two chambers, and the transepithelial flux of a high molecular weight protein is measured by labeling the molecule with a fluorescent dye.

CONTACTS AND LOCATIONS:
Locations (1):
- Jan Tack, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided